CLINICAL TRIAL: NCT01651975
Title: Evaluation of Two Different Thickening Products in Patients With Dysphagia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 200917127
Record Dates: First submitted 2012-01-24; First posted 2012-07-27 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Dysphagia
Keywords: Dysphagia; Thickening liquid; Thickening agent; Fluoroscopic swallow study; Aspiration; History of dysphagia; DSS; Age > 18; comprehensive DSS; informed consent
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thickenup (Other)
  Interventions: Dietary Supplement: Thickenup; Dietary Supplement: Thickenup Advance

INTERVENTIONS:
Dietary Supplement: Thickenup — given two 1-cc boluses of liquid contrast agent (barium), one 3-cc of thin liquid contrast, one 3-cc of paste, one cookie with contrast, one 20-cc bolus of liquid contrast, and one 20-cc bolus of thin liquid contrast. The patients are then studied in the anterior/posterior view with one 1-cc, one 3-cc, and one 20-cc bolus of thin liquid barium 1-4. At the end of the protocol patients are routinely administered products with either starch or gel based thickener to evaluate the swallowing safety of the thickened agent. The protocol includes a 3-minute limitation on total fluoroscopy time to ensure clinician and patient safety.
  Other Names: Liquid E-Z-Paque; E-Z-Em, Inc.
Dietary Supplement: Thickenup Advance — given two 1-cc boluses of liquid contrast agent (barium), one 3-cc of thin liquid contrast, one 3-cc of paste, one cookie with contrast, one 20-cc bolus of liquid contrast, and one 20-cc bolus of thin liquid contrast. The patients are then studied in the anterior/posterior view with one 1-cc, one 3-cc, and one 20-cc bolus of thin liquid barium 1-4. At the end of the protocol patients are routinely administered products with either starch or gel based thickener to evaluate the swallowing safety of the thickened agent. The protocol includes a 3-minute limitation on total fluoroscopy time to ensure clinician and patient safety.
  Other Names: Liquid E-Z Paque; E-Z-EM, Inc

SUMMARY:
Dysphagia is extremely common. The importance of providing adequate nutritional support to persons with dysphagia is the cornerstone to exceptional care. Diet modification with thickening agents is an essential aspect of this nutritional support. The purpose of this investigation is to compare the efficacy of a starch based (Thickenup or TU) to a gel based thickening agent (Thickenup Advance or TUA).

DETAILED DESCRIPTION:
Swallowing problems (dysphagia) are encountered frequently in primary practice and in the hospital setting. The list of possible causes is large, ranging from strokes and neurological disease to complications of cancer treatment, acid reflux, and surgery. Many patients have a reduced ability to feel food and fluid (reduced sensation) within the throat (pharynx) and this leads to an inability to manipulate food and fluids in the correct manner. This can produce a variety of swallowing problems such as choking on foods and fluids, regurgitation, aspiration, weight loss, malnutrition and poor quality of life.

Treatment of dysphagia is largely directed at rehabilitation of muscle power and education about safe swallowing techniques or positioning that limits food and fluid from entering the airway. One of the most widely accepted treatments of dysphagia is to alter the texture of food. Most patients with dysphagia will have more difficulty swallowing thin liquids. By adding a thickener to the liquid, a food bolus becomes more cohesive, and is less likely to become aspirated. Various types of thickening products are available over-the-counter without a prescription. These thickening products are bland and currently have no flavor. The investigators hypothesize that alterations in food taste (sweet, salty, etc…), viscosity will improve swallowing efficiency. The purpose of this investigation is to evaluate the effects of food taste, texture on swallowing efficiency. The goal is to develop safer, better tasting food products and improve the quality of life in patients with disabling swallowing disorders.

ELIGIBILITY:
Inclusion Criteria:

* History of dysphagia necessitating a dynamic fluoroscopic swallow study
* Age > 18 years
* Ability to complete a comprehensive dynamic fluoroscopic swallow study
* Ability to provide informed consent for study participation

Exclusion Criteria:

* Age < 18 years
* Pregnant women
* Prisoner or other institutionalized individual
* Cognitive disability precluding the ability to provide informed consent or complete a comprehensive swallow study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Compare aspiration risk | Time of intervention
  Compare the prevalence of aspiration risk with TUA to the prevalence of aspiration risk with TU and thin liquid barium at the time the subject undergoes a fluoroscopic swallowing study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Belafsky, MD, Ph.D., Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Medical Center, Sacramento, California, United States